CLINICAL TRIAL: NCT04132531
Title: Impact of Bariatric Surgery on Circulating Inflammatory and Pro-vascular Progenitor Cell Populations.
Brief Title: Effect of Weight Loss Surgery on Stem Cells.
Status: Completed | Type: Observational
Sponsor: Unity Health Toronto (Other)
Collaborators: Humber River Hospital (Other); University of Western Ontario, Canada (Other)
Responsible Party: Principal Investigator, Subodh Verma, Clinical Professor of Surgery and Pharmacology & Toxicology, Unity Health Toronto
Other Study IDs: PRO_B_001
Record Dates: First submitted 2019-10-10; First posted 2019-10-18 (Actual); Last update posted 2019-10-18 (Actual); Status verified 2019-10

CONDITIONS: Obesity, Morbid; Stem Cells; Cardiovascular Morbidity
Keywords: Stem Cells; Obesity; Cardiovascular Events; Type 2 Diabetes
MeSH Terms: conditions — Obesity, Morbid; Obesity; Diabetes Mellitus, Type 2 | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum was collected and stored.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Normal weight control: Individuals who are generally healthy and have a body mass index less than 25 kg/m^2.
- Bariatric Surgery Group: Individuals electing to undergo bariatric surgery (generally with a body mass index between 35 and 40 kg/m^2 with an additional co-morbidity such as type 2 diabetes, or individuals with a body mass index greater than 40 kg/m^2) and who are willing to participate for 2 visits, one before and one after surgery. The intervention in this group is bariatric surgery.
  Interventions: Procedure: Bariatric (weight loss) surgery

INTERVENTIONS:
Procedure: Bariatric (weight loss) surgery — Surgical intervention for weight reduction, whereby the stomach is resected and the gastrointestinal tract is rerouted in the case of Roux-en-y gastric bypass, or the stomach is only resected in the case of sleeve gastrectomy.
  Groups: Bariatric Surgery Group

SUMMARY:
Obesity and diabetes are linked to increased risk for health problems such as heart attack, stroke, and death. At the cellular level, obesity and diabetes increase levels of harmful inflammatory cells (M1 macrophages) and decreases levels of protective stem cells (circulating progenitor cells) in the blood.

Bariatric (weight loss) surgery is an effective treatment that leads to significant weight loss and improved health in patients with obesity. However, it is unknown if weight loss surgery also replenishes healthy stem cells and decreases inflammatory cells in the body. Therefore, the purpose of this research study is to compare levels of these stem and inflammatory cells before and after bariatric surgery, and to compare to a control group of healthy normal weight participants.

The investigators anticipate that inflammatory cell levels will be reduced and stem cell levels and function will be restored after bariatric surgery, similar to levels of healthy normal weight individuals.

DETAILED DESCRIPTION:
The escalating pandemics of obesity and type 2 diabetes mellitus (T2DM) are among the most devastating health crises worldwide. The prevalence of obesity (body mass index (BMI) > 30kg/m^2) is nearly 1 billion individuals worldwide and estimated by the Center for Disease Control at 37.7 percent of the adult population in the United States. The International Diabetes Federation estimates that over 400 million individuals worldwide have T2DM and this number is expected to increase to over 600 million by the year 2040. Diet, exercise, and medications such as metformin have long been the cornerstone of T2DM therapy. Unfortunately, long-term success in the control of T2DM remain disappointing, and even with new medications such as glucagon-like peptide-1 (GLP-1) analogues (Liraglutide) and sodium-glucose co-transporter 2 (SGLT2) inhibitors (Gliflozins), adequate glycemic control remains elusive. Ultimately, T2DM patients will develop severe cardiovascular complications such as peripheral artery disease, heart attack, and stroke. Due to aging population demographics, and the paucity of curative therapies in this area, the prevalence and economic burden of obesity and T2DM is on the rise. Currently, the costs of medical care for obesity-related illnesses in the United States are estimated at $147 - 185 billion per year. Therefore, the search for curative therapies to combat obesity and T2DM are continually sought.

Bariatric surgery is increasingly recognized as one of the most effective interventions to help patients achieve significant and sustained weight loss, and improved metabolic health. Permanent loss of 20-25 percent body weight (35 - 45 kilograms) is common for patients receiving Roux-en-y Gastric Bypass (RYGB) or Vertical Sleeve Gastrectomy (VSG) compared to <5 percent in best non-surgical medical therapy patients. The mechanisms of weight loss following bariatric surgery are multifactorial and include changes in food intake, satiety, alterations in gut hormones and bile acid adaptations. Such drastic weight loss is also associated with improvement in chronic inflammatory diseases, including atherosclerosis and T2DM. Indeed, bariatric surgery leads to improved glycemic control and potential remission of T2DM. Recently, studies have independently reported significant reductions in fasting blood glucose and glycated hemoglobin (HbA1C) in >80 percent of patients receiving bariatric surgery. Amelioration of T2DM commonly occurs within days to weeks of surgery even before substantial weight loss is observed. Finally, adverse cardiovascular events, usually associated with obesity and T2DM, were reduced after bariatric surgery compared to conventional therapies. Despite these phenomenal successes, the mechanisms governing the reversal of diabetes after bariatric surgery remains largely unknown.

Obesity, atherosclerotic plaque formation and the development of T2DM are all associated with heightened inflammation. Obesity involves increases in inflammatory immune cells (M1 macrophages) that are present during the remodeling of adipose tissue. In functional opposition to heightened immunity is the reparative role of tissue-specific stem cells. Central to all regenerative processes, stem cells can be found within every tissue in the body with the capacity to self-renew, and to generate new cell types that promote tissue maintenance or repair. In this capacity, stem cells can be considered "conductors of the orchestra" that co-ordinate the myriad cells and signals involved in the regenerative response. However, during chronic diseases such as T2DM, relentless inflammation and oxidative damage results in stem cell depletion and dysfunction, and the severity of injury overwhelms the capacity to respond. For example, adipose tissue contains a heterogenous mixture of stem and progenitor cells which are likely affected by the inflammation associated with obesity. Similarly, circulating hematopoietic and endothelial progenitor cells, involved in blood vessel maintenance and repair, show aberrant secretory and vessel formative functions that are negatively impacted by chronic hyperlipidemia and hyperglycemia. This concept termed "stem cell exhaustion" is becoming increasingly recognized during chronic diseases, as circulating stem and progenitor cell number and/or regenerative function is altered by the inflammatory environment within obesity/T2DM patients.

What remains unclear is whether reduced circulating stem cell number or aberrant regenerative function can be restored following bariatric surgery. The investigators have recently established novel methodologies to assess inflammatory status (M1 / M2 macrophage status) and circulating progenitor cell content and function by performing detailed flow cytometric analyses using aldehyde dehydrogenase (ALDH, a detoxification enzyme and conserved stem cell function) in combination with cell surface marker analyses. Notably, the investigators have shown that circulating progenitor cell content and inflammatory M1 macrophage content are increased in patients with T2DM compared to age-matched healthy controls. For the first time, the effectiveness of bariatric surgery at the cellular level can be evaluated and regenerative stem cell functions that impact obesity and T2DM can be explored. Elucidating the status of stem cells following bariatric surgery will provide insight into the likelihood of T2DM relapse or reverting to an obese state and provide a potential mechanism for the improvements in cardiovascular health. This study will be able to establish a relationship between the reversal of obesity, T2DM and adverse cardiovascular events with the restoration of regenerative stem cell associated with anti-inflammatory and pro-angiogenic function.

The investigators hypothesize that bariatric surgery will augment circulating, pro-vascular progenitor cell content and will reduce systemic inflammation via restoration of M1 / M2 macrophage balance.

ELIGIBILITY:
Inclusion Criteria:

* Individuals undergoing bariatric surgery
* Must be able to provide two visits, before and after surgery

Exclusion Criteria:

* Unable to provide written consent
* Unable to provide two visits for blood collection

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Community Sample/Residents mainly from the Greater Toronto Area.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-06-25 (Actual); Study Completion 2019-08-13 (Actual)

PRIMARY OUTCOMES:
Change in the frequency of circulating cells with aldehyde dehydrogenase activity. | Baseline and after surgery, 3-4 months

SECONDARY OUTCOMES:
Change in the frequency of circulating cells with aldehyde dehydrogenase activity and cell surface marker expression. | Baseline and after surgery, 3-4 months

OTHER OUTCOMES:
Changes in the concentration of oxidative stress and inflammatory markers | Baseline and after surgery, 3-4 months

CONTACTS AND LOCATIONS:
Overall Officials: Subodh Verma, MD, Principal Investigator — Unity Health Toronto; David A Hess, PhD, Principal Investigator — Robart's Research Institute, London, Ontario
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, ICF
Time Frame: Starting 6 month following publication.

REFERENCES:
- [Background] Kahn SE, Hull RL, Utzschneider KM. Mechanisms linking obesity to insulin resistance and type 2 diabetes. Nature. 2006 Dec 14;444(7121):840-6. doi: 10.1038/nature05482. PMID 17167471
- [Background] Adler BJ, Kaushansky K, Rubin CT. Obesity-driven disruption of haematopoiesis and the bone marrow niche. Nat Rev Endocrinol. 2014 Dec;10(12):737-48. doi: 10.1038/nrendo.2014.169. Epub 2014 Oct 14. PMID 25311396
- [Background] Benites BD, Gilli SC, Saad ST. Obesity and inflammation and the effect on the hematopoietic system. Rev Bras Hematol Hemoter. 2014 Mar;36(2):147-51. doi: 10.5581/1516-8484.20140032. PMID 24790541
- [Background] Forsythe LK, Wallace JM, Livingstone MB. Obesity and inflammation: the effects of weight loss. Nutr Res Rev. 2008 Dec;21(2):117-33. doi: 10.1017/S0954422408138732. PMID 19087366
- [Background] Flegal KM, Kruszon-Moran D, Carroll MD, Fryar CD, Ogden CL. Trends in Obesity Among Adults in the United States, 2005 to 2014. JAMA. 2016 Jun 7;315(21):2284-91. doi: 10.1001/jama.2016.6458. PMID 27272580
- [Background] Stirban AO, Tschoepe D. Cardiovascular complications in diabetes: targets and interventions. Diabetes Care. 2008 Feb;31 Suppl 2:S215-21. doi: 10.2337/dc08-s257. PMID 18227488
- [Background] Cawley J, Meyerhoefer C. The medical care costs of obesity: an instrumental variables approach. J Health Econ. 2012 Jan;31(1):219-30. doi: 10.1016/j.jhealeco.2011.10.003. Epub 2011 Oct 20. PMID 22094013
- [Background] Finkelstein EA, Trogdon JG, Cohen JW, Dietz W. Annual medical spending attributable to obesity: payer-and service-specific estimates. Health Aff (Millwood). 2009 Sep-Oct;28(5):w822-31. doi: 10.1377/hlthaff.28.5.w822. Epub 2009 Jul 27. PMID 19635784
- [Background] Keidar A. Bariatric surgery for type 2 diabetes reversal: the risks. Diabetes Care. 2011 May;34 Suppl 2(Suppl 2):S361-266. doi: 10.2337/dc11-s254. No abstract available. PMID 21525483
- [Background] Kashyap SR, Gatmaitan P, Brethauer S, Schauer P. Bariatric surgery for type 2 diabetes: weighing the impact for obese patients. Cleve Clin J Med. 2010 Jul;77(7):468-76. doi: 10.3949/ccjm.77a.09135. PMID 20601620
- [Background] Ponce J, Nguyen NT, Hutter M, Sudan R, Morton JM. American Society for Metabolic and Bariatric Surgery estimation of bariatric surgery procedures in the United States, 2011-2014. Surg Obes Relat Dis. 2015 Nov-Dec;11(6):1199-200. doi: 10.1016/j.soard.2015.08.496. Epub 2015 Aug 12. No abstract available. PMID 26476493
- [Background] Ponce J, DeMaria EJ, Nguyen NT, Hutter M, Sudan R, Morton JM. American Society for Metabolic and Bariatric Surgery estimation of bariatric surgery procedures in 2015 and surgeon workforce in the United States. Surg Obes Relat Dis. 2016 Nov;12(9):1637-1639. doi: 10.1016/j.soard.2016.08.488. Epub 2016 Aug 26. No abstract available. PMID 27692915
- [Background] Khan S, Rock K, Baskara A, Qu W, Nazzal M, Ortiz J. Trends in bariatric surgery from 2008 to 2012. Am J Surg. 2016 Jun;211(6):1041-6. doi: 10.1016/j.amjsurg.2015.10.012. Epub 2015 Dec 11. PMID 26762828
- [Background] Schauer PR, Bhatt DL, Kirwan JP, Wolski K, Aminian A, Brethauer SA, Navaneethan SD, Singh RP, Pothier CE, Nissen SE, Kashyap SR; STAMPEDE Investigators. Bariatric Surgery versus Intensive Medical Therapy for Diabetes - 5-Year Outcomes. N Engl J Med. 2017 Feb 16;376(7):641-651. doi: 10.1056/NEJMoa1600869. PMID 28199805
- [Background] Mulla CM, Middelbeek RJW, Patti ME. Mechanisms of weight loss and improved metabolism following bariatric surgery. Ann N Y Acad Sci. 2018 Jan;1411(1):53-64. doi: 10.1111/nyas.13409. Epub 2017 Sep 3. PMID 28868615
- [Background] Baptista LS, Silva KR, Borojevic R. Obesity and weight loss could alter the properties of adipose stem cells? World J Stem Cells. 2015 Jan 26;7(1):165-73. doi: 10.4252/wjsc.v7.i1.165. PMID 25621116
- [Background] Adams TD, Davidson LE, Litwin SE, Kim J, Kolotkin RL, Nanjee MN, Gutierrez JM, Frogley SJ, Ibele AR, Brinton EA, Hopkins PN, McKinlay R, Simper SC, Hunt SC. Weight and Metabolic Outcomes 12 Years after Gastric Bypass. N Engl J Med. 2017 Sep 21;377(12):1143-1155. doi: 10.1056/NEJMoa1700459. PMID 28930514
- [Background] Pories WJ, Swanson MS, MacDonald KG, Long SB, Morris PG, Brown BM, Barakat HA, deRamon RA, Israel G, Dolezal JM, et al. Who would have thought it? An operation proves to be the most effective therapy for adult-onset diabetes mellitus. Ann Surg. 1995 Sep;222(3):339-50; discussion 350-2. doi: 10.1097/00000658-199509000-00011. PMID 7677463
- [Background] Schauer PR, Burguera B, Ikramuddin S, Cottam D, Gourash W, Hamad G, Eid GM, Mattar S, Ramanathan R, Barinas-Mitchel E, Rao RH, Kuller L, Kelley D. Effect of laparoscopic Roux-en Y gastric bypass on type 2 diabetes mellitus. Ann Surg. 2003 Oct;238(4):467-84; discussion 84-5. doi: 10.1097/01.sla.0000089851.41115.1b. PMID 14530719
- [Background] Romeo S, Maglio C, Burza MA, Pirazzi C, Sjoholm K, Jacobson P, Svensson PA, Peltonen M, Sjostrom L, Carlsson LM. Cardiovascular events after bariatric surgery in obese subjects with type 2 diabetes. Diabetes Care. 2012 Dec;35(12):2613-7. doi: 10.2337/dc12-0193. Epub 2012 Aug 1. PMID 22855732
- [Background] Sjostrom L, Peltonen M, Jacobson P, Sjostrom CD, Karason K, Wedel H, Ahlin S, Anveden A, Bengtsson C, Bergmark G, Bouchard C, Carlsson B, Dahlgren S, Karlsson J, Lindroos AK, Lonroth H, Narbro K, Naslund I, Olbers T, Svensson PA, Carlsson LM. Bariatric surgery and long-term cardiovascular events. JAMA. 2012 Jan 4;307(1):56-65. doi: 10.1001/jama.2011.1914. PMID 22215166
- [Background] Mathieu P, Lemieux I, Despres JP. Obesity, inflammation, and cardiovascular risk. Clin Pharmacol Ther. 2010 Apr;87(4):407-16. doi: 10.1038/clpt.2009.311. Epub 2010 Mar 3. PMID 20200516
- [Background] Kizil C, Kyritsis N, Brand M. Effects of inflammation on stem cells: together they strive? EMBO Rep. 2015 Apr;16(4):416-26. doi: 10.15252/embr.201439702. Epub 2015 Mar 4. PMID 25739812
- [Background] Oh J, Lee YD, Wagers AJ. Stem cell aging: mechanisms, regulators and therapeutic opportunities. Nat Med. 2014 Aug;20(8):870-80. doi: 10.1038/nm.3651. PMID 25100532
- [Background] El-Tantawy WH, Haleem EN. Therapeutic effects of stem cell on hyperglycemia, hyperlipidemia, and oxidative stress in alloxan-treated rats. Mol Cell Biochem. 2014 Jun;391(1-2):193-200. doi: 10.1007/s11010-014-2002-x. Epub 2014 Mar 7. PMID 24604673
- [Background] Wu CL, Diekman BO, Jain D, Guilak F. Diet-induced obesity alters the differentiation potential of stem cells isolated from bone marrow, adipose tissue and infrapatellar fat pad: the effects of free fatty acids. Int J Obes (Lond). 2013 Aug;37(8):1079-87. doi: 10.1038/ijo.2012.171. Epub 2012 Nov 20. PMID 23164698
- [Result] Sherman SE, Kuljanin M, Cooper TT, Putman DM, Lajoie GA, Hess DA. High Aldehyde Dehydrogenase Activity Identifies a Subset of Human Mesenchymal Stromal Cells with Vascular Regenerative Potential. Stem Cells. 2017 Jun;35(6):1542-1553. doi: 10.1002/stem.2612. Epub 2017 Apr 3. PMID 28295901
- [Result] Jialal I, Devaraj S, Singh U, Huet BA. Decreased number and impaired functionality of endothelial progenitor cells in subjects with metabolic syndrome: implications for increased cardiovascular risk. Atherosclerosis. 2010 Jul;211(1):297-302. doi: 10.1016/j.atherosclerosis.2010.01.036. Epub 2010 Feb 4. PMID 20171637
- [Result] Seneviratne AK, Bell GI, Sherman SE, Cooper TT, Putman DM, Hess DA. Expanded Hematopoietic Progenitor Cells Reselected for High Aldehyde Dehydrogenase Activity Demonstrate Islet Regenerative Functions. Stem Cells. 2016 Apr;34(4):873-87. doi: 10.1002/stem.2268. Epub 2016 Jan 19. PMID 26676482
- [Derived] Hess DA, Trac JZ, Glazer SA, Terenzi DC, Quan A, Teoh H, Al-Omran M, Bhatt DL, Mazer CD, Rotstein OD, Verma S. Vascular Risk Reduction in Obesity through Reduced Granulocyte Burden and Improved Angiogenic Monocyte Content following Bariatric Surgery. Cell Rep Med. 2020 May 19;1(2):100018. doi: 10.1016/j.xcrm.2020.100018. eCollection 2020 May 19. PMID 33205058